CLINICAL TRIAL: NCT05487391
Title: QL1706 Combined With Platinum-based Chemotherapy Versus Placebo Combined With Platinum-based Chemotherapy as Adjuvant Therapy for Stage II-IIIB Non-small Cell Lung Cancer After Complete Surgical Resection: a Randomized, Double-blind, Multicenter Phase III Clinical Study.
Brief Title: A Study of QL1706 Combined With Platinum-containing Chemotherapy in Adjuvant Treatment of Stage II-IIIB Non-small Cell Lung Cancer After Complete Surgical Resection.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL1706-304
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Paclitaxel; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 plus Platinum-based chemotherapy (Experimental): QL1706(5mg/kg Q3W IV) plus Platinum-based chemotherapy
  Interventions: Drug: QL1706 injection; Drug: Vinorelbine Tartrate; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Placebo plus Platinum-based chemotherapy (Placebo Comparator): Placebo(5mg/kg Q3W IV) plus Platinum-based chemotherapy
  Interventions: Drug: Vinorelbine Tartrate; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Placebo

INTERVENTIONS:
Drug: QL1706 injection — QL1706(5mg/kg Q3W IV) concomitantly with Platinum-based chemotherapy
  Arms: QL1706 plus Platinum-based chemotherapy
Drug: Vinorelbine Tartrate — Vinorelbine 25mg/m2（D1、D8）Q3W IV, 2-4 cycles
Drug: Paclitaxel — Paclitaxel 175mg/m2（D1） Q3W IV, 2-4 cycles
Drug: Cisplatin — Cisplatin 75mg/m2（D1）Q3W IV, 2-4 cycles
Drug: Carboplatin — Carboplatin AUC=5（D1） Q3W IV, 2-4 cycles
Drug: Pemetrexed — Pemetrexed 500mg/m2（D1） Q3W IV, 2-4 cycles
Drug: Placebo — Placebo
  Arms: Placebo plus Platinum-based chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of QL1706 combined with platinum-based chemotherapy versus placebo combined with platinum-based chemotherapy in adjuvant treatment of stage II-IIIB NSCLC without EGFR-sensitizing mutations and ALK fusions after complete surgical resection.The subjects were randomly divided into two groups according to 1:1, with about 316 subjects in the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participated, signed an informed consent form (ICF), and were able to follow the study procedures.
* Histopathologically confirmed squamous or non-squamous non-small cell lung cancer
* Stage II-IIIB according to the 8th edition of the American Joint Committee on Cancer (AJCC) , and had received radical surgical resection (R0) treatment.
* Participants were enrolled to receive adjuvant therapy within 10 weeks after surgery (≤70 days) and had to recover sufficiently from surgery.
* Non-squamous NSCLC subjects without EGFR-sensitizing mutation or ALK fusion gene.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subjects (including women and men) agreed to use effective contraception from the time of signing the informed consent to 180 days after the last use of the study drug.

Exclusion Criteria:

* Currently participating in and receiving study treatment or participating in an investigational drug study and receiving study treatment or using an investigational device within 4 weeks prior to the first dose of study treatment.
* Previous treatment with neoadjuvant/adjuvant chemotherapy or immune checkpoint inhibitor therapy.
* Cardiovascular and cerebrovascular diseases with clinical significance.
* Gastrointestinal disease of clinical significance.
* Clinically significant lung damage.
* Human immunodeficiency virus (HIV) antibody positive; Treponema pallidum antibody positive.
* Active uncontrolled hepatitis B or active hepatitis C.
* Administer a live vaccine within 30 days prior to the first dose of study treatment.
* Other malignancies occurred within 5 years prior to study enrollment. (Except: Bowen's disease; cured basal cell or squamous cell skin cancer; prostate cancer with a Gleason score of 6; treated cervical carcinoma in situ.)
* Previously allergic to macromolecular protein preparations, or to any component of QL1706 and other investigational drugs; history of severe allergy to chemotherapy drugs (pemetrexed, vinorelbine, paclitaxel, cisplatin, carboplatin) or their preventive drugs, etc.
* History of psychotropic substance abuse, alcohol or drug abuse; prior history of clear neurological or psychiatric disorders, including epilepsy or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-05-22 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) in the PD-L1 ≥1% Population, Assessed by Investigator. | Up to approximately 84 months
  DFS was defined as the time from randomization to first recurrence of NSCLC, appearance of new primary NSCLC, or death from any cause, whichever occurred first. Tumor recurrence includes local recurrence and distant metastasis.
Disease-free Survival (DFS) in the ITT Population, Assessed by Investigator. | Up to approximately 84 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 108 months
  OS is defined as the time from random to death from any cause. OS will be measured in the PD-L1 subpopulation and in the ITT population.
Percentage of Participants Who are Survival at Year 4 | Year 4
  OS rates will be measured in the PD-L1 subpopulation and in the ITT population.
Percentage of Participants Who are Disease-Free at Year 3 | Year 3
  DFS rates will be measured in the PD-L1 subpopulation and in the ITT population.
Percentage of Participants Who are Disease-Free at Year 5 | Year 5
  DFS rates will be measured in the PD-L1 subpopulation and in the ITT population.
DFS Within Selected Populations | Up to approximately 108 months
  Assessed by Investigator
Percentage of Participants with Adverse Events and Serious Adverse Events | Up to approximately 108 months

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, PhD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai. China, Shanghai, China

REFERENCES:
- [Derived] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938